CLINICAL TRIAL: NCT02599454
Title: A Phase I Trial of an Immune Checkpoint Inhibitor Plus Stereotactic Ablative Radiotherapy in Patients With Inoperable Stage I Non-Small Cell Lung Cancer
Brief Title: Atezolizumab and Stereotactic Body Radiation Therapy in Treating Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Megan Daly, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Megan Daly, MD, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 774542; UCDCC#258 (Other: UC Davis); ML29955 (Other Grant/Funding Number: Genentech); UCDCC#258 (Other: University of California Davis Comprehensive Cancer Center); NCI-2015-01796 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Stage I Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- atezolizumab + SBRT (Experimental): DOSE ESCALATION PHASE: Patients receive atezolizumab IV over 30-60 minutes on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Within 24-48 hours after receiving atezolizumab, patients also undergo 4-5 fractions of stereotactic body radiation therapy over days 1-5 of course 3.
  EXPANSION PHASE: Patients receive atezolizumab IV over 30-60 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Within 24-48 hours after receiving atezolizumab, patients also undergo 4-5 fractions of stereotactic body radiation therapy over days 1-5 of course 3.
  Interventions: Drug: Atezolizumab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Atezolizumab — Into the vein Day 1 every 3 weeks for 6 cycles
  Other Names: MPDL3280A
Radiation: Stereotactic Body Radiation Therapy — Radiation therapy will be performed to 50 Gy over 4 fractions of 12/5 Gy each for peripherally located tumors and 50 Gy over 5 fractions of 10 Gy each for centrally located tumors
  Other Names: SBRT

SUMMARY:
This phase I trial studies the side effects and best dose of atezolizumab that can be given together with stereotactic body radiation therapy (SBRT) in treating patients with stage I non-small cell lung cancer that cannot be removed by surgery. Monoclonal antibodies, such as atezolizumab, may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Stereotactic body radiation therapy is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may kill more tumor cells and cause less damage to normal tissue. Giving atezolizumab together with stereotactic body radiation therapy may kill more tumor cells and be a better treatment for non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of MPDL3280A (atezolizumab) that can be given with stereotactic ablative radiotherapy (SAR) (stereotactic body radiation therapy) in patients with inoperable stage I non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To characterize the safety profile of this regimen using CTCAE v4 (Common Toxicity Criteria for Adverse Events version 4).

II. To provide preliminary efficacy data of the combination as determine by objective response rate and disease free survival using RECIST 1.1 (Response Evaluation Criteria for Solid Tumors) and Immune Related RECIST (irRECIST).

TERTIARY OBJECTIVES:

I. To analyze serial blood for change in cytokine signatures, fluorescence activated cell sorting (FACS) and immunophenotyping of peripheral blood mononuclear cells (PBMCs) and tumor infiltrating immune cells.

II. To evaluate pre and post treatment tumor tissue (if available) for programmed cell death-ligand 1 (PD-L1) and other immune proteins in the tumor and tumor microenvironment and for molecular profiling in a subset of patient samples.

III. To discover biomarkers of response from the data obtained.

OUTLINE: This is a dose-escalation study of atezolizumab.

DOSE ESCALATION PHASE: Patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Within 24-48 hours after receiving atezolizumab, patients also undergo 4-5 fractions of stereotactic body radiation therapy over days 1-5 of course 3.

EXPANSION PHASE: Patients receive atezolizumab IV over 30-60 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Within 24-48 hours after receiving atezolizumab, patients also undergo 4-5 fractions of stereotactic body radiation therapy over days 1-5 of course 3.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven stage I NSCLC =< 5 cm diameter
* One or more high-risk features identified:

  * Tumor diameter >= 2 cm
  * Tumor standardized uptake value maximum (SUVmax) >= 6.2
  * Moderately, poorly differentiated or undifferentiated histology
* Evaluable disease per RECIST 1.1
* Patients must be medically or surgically inoperable as determined by a physician OR unwilling to undergo surgical resection
* All patients must have an forced expiratory volume in 1 second (FEV1) >= 700cc
* All patients must have a carbon monoxide diffusing capability test (DLCO) >= 5.5 m/min/mmHg
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2
* Life expectancy >= 12 months
* Absolute neutrophil count (ANC) > 1500 cells/uL
* White blood cell count (WBC) > 2500/uL
* Lymphocyte count > 500/uL
* Platelet count > 100,000/uL
* Hemoglobin > 9 g/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN) with alkaline phosphatase =< 2.5 x ULN OR AST and ALT =< 1.5 x ULN, with alkaline phosphatase > 2.5 x ULN
* Serum bilirubin =< 1.0 x ULN
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) < 1.5 x ULN (for patients on anticoagulation they must be receiving a stable dose for at least 1 week prior to enrollment)
* Creatinine clearance > 30 mL/min by Cockcroft-Gault formula
* No history of severe hypersensitivity reactions to other monoclonal antibodies (mAbs)
* No other active malignancy
* Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible
* Patients with controlled type 1 diabetes mellitus on a stable insulin regimen are eligible
* Archival tumor sample available; tissue from an fine-needle aspiration (FNA) is allowed but tumor tissue from a core needle biopsy is preferred
* For female patients of childbearing potential and male patients with partners of childbearing potential agreement (by patient and/or partner) to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [< 1% per year] when used consistently and correctly) and to continue its use for 6 months after the last dose of MPDL3280A
* Signed informed consent
* Ability to comply with the protocol

Exclusion Criteria:

* Uncontrolled concomitant disease
* Significant cardiovascular disease (New York Heart Association Class [NYHA] class II or greater); myocardial infarction within 3 month prior to randomization, unstable arrhythmias, unstable angina or a patient with a known left ventricular ejection fraction (LVEF) < 40%
* Severe infection within 4 weeks prior to enrollment
* Active tuberculosis
* Oral or IV antibiotics within 2 weeks or 5 half-lives prior to enrollment
* History of autoimmune disease
* Positive for human immunodeficiency virus (HIV), hepatitis B (hepatitis B surface antigen [HBsAg] reactive), or hepatitis C virus (hepatitis C virus ribonucleic acid [HCV RNA] [qualitative] is detected)
* History of idiopathic pulmonary fibrosis, drug-induced pneumonitis, organizing pneumonia
* Treatment with systemic immunostimulatory agents within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrollment
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications within past 4 weeks or 5 half-lives whichever is shorter
* Pregnant and/or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 9 weeks
  The adverse events will be summarized as frequency, proportion of patients MTD. The exact 95% confidence interval for proportion will be categorized by type, severity, nadir or maximum values for the laboratory measures, time of onset, duration, and reversibility or outcome. Tables will be created to summarize these toxicities by dose and course.

SECONDARY OUTCOMES:
Disease free survival (DFS), assessed by RECIST 1.1 and irRECIST | Up to 5 years
  DFS will be summarized with Kaplan-Meier plots. The median DFS time will be estimated using standard life table methods.
Overall response rate (ORR), assessed by RECIST 1.1 | Time from the start of the treatment until disease progression/recurrence, assessed up to 5 years
  ORR will be summarized by exact binomial confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kelly, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - David Grant United States Air Force Medical Center, Travis AFB, California

IPD SHARING:
Plan to Share IPD: No